CLINICAL TRIAL: NCT04878796
Title: Observational Study to Monitor the Effects of the COVID-19 Vaccine on Cancer Patients Receiving Active Therapy (ANTICOV).
Brief Title: Effectiveness of mRNA Covid-19 Vaccines on Cancer Patients:Observational Study. (ANTICOV)
Acronym: ANTICOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale di Cremona (Other)
Responsible Party: Sponsor
Other Study IDs: ASST CR-01-2021
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-05

CONDITIONS: Cancer; Covid-19; Vaccine Response
Keywords: Cancer treatment; Covid-19; Vaccine
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum collection, adverse events collection — Measuring Abs variation at different timepoints compared to baseline. LIAISON SARS-Cov-2 TrimericS IgG and Elecsys anti-SARS-Cov-2 tests will be adopted. The level of Abs will be evaluated at baseline and 30(±7), 180(±7),365(±7)days after the 2nd dose of vaccine

SUMMARY:
Based on recent data, COVID (COV) vaccination in cancer patients (pts) is strictly recommended. For oncologic pts,2 types of m-RNA vaccines have been approved: BNT162b2 (Pfizer, Biontech) and mRNA-1273 (Moderna, NIAID). In immunocompetent population, the administration of 2 doses confers 95% protection against COV. However, protection conferred by vaccines, adverse events (AEs) and correlations with antiblastic treatments are unknown in cancer pts.

DETAILED DESCRIPTION:
Trial Design

This is a monocentric observational study conducted by the Oncology Unit of Cremona (CR) Hospital, enrolling pts from Oncology, Hematology, Radiotherapy and Palliative Care of Cr Hospital.

This trial aims to prospectively and retrospectively evaluate the effectiveness of mRNA vaccines [BNT162b2 (Pfizer) and mRNA-1273 (Moderna)], the quantization of the antibodies (Abs) response and the onset of AEs in a consecutive population of 300 cancer pts, undergoing antiblastic treatment, starting from March 26Th,2021.

From March, 2021 a vaccination point was set up by Cr Hospital, specific for cancer pts. Vaccine is administered at least 5 days after the last dose of intravenous or oral chemotherapy treatment; the next course of therapy is not administered within the next 3 days. Target therapy and immunotherapy doesn't need interruptions.

- Primary endpoint: Evaluating the protection conferred by vaccination, by detecting the number of symptomatic pts affected by COV, diagnosed 7-60 days after the 2nddose of vaccine. Confirmed of COV infection is defined according to the Food and Drug Administration criteria combined with a nasopharyngeal swab, positive for SARS-Cov-2, obtained during the symptomatic period or within 4 days before or after it.

- Secondary endpoints: Measuring Abs variation at different timepoints compared to baseline. LIAISON SARS-Cov-2 TrimericS IgG and Elecsys anti-SARS-Cov-2 tests will be adopted. The level of Abs will be evaluated at baseline and 30(±7), 180(±7),365(±7)days after the 2nd dose of vaccine;

Describing AEs; Evaluating the interference between vaccine and cancer treatments; Analysis of the Abs subtypes; Duration of abs, up to 12 months after 2nd dose

Statistic Analysis The hypothesis of vaccine inferiority in the trial population is rejected if a rate of protection conferred by the vaccine is observed in 89% of the sample size. The null hypothesis will be rejected if out of a sample size of 300 patients at least 261 are "protected".

The observed proportion of patients with protection will be described by absolute and relative frequency, with Clopper-Pearson confidence intervals. The primary objective will be tested by non-inferiority one-single proportion test, compared with the historical value of 95%. In order to describe the trend of antibody changes in the multiple detections, the ANOVA test for repeated measurements will be used.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients receiving active therapy (chemotherapy, immunotherapy, target therapy, radiotherapy)
* Cancer patients receiving hormonal therapy for metastatic disease.
* Must be ≥18 years of age.
* Written, signed consent for study participation.

Exclusion Criteria:

* Cancer patients receiving hormonal therapy in adjuvant regimen.
* Patients in follow-up and who have completed their cancer treatment for > 6 months.
* Life expectancy less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients receiving active therapy (chemotherapy, immonotherapy, target therapy, radiotherapy, hormonal therapy ) or who have completed their oncologic treatment within 6 months and have been prescribed the administration of the admRNAanti-COVID-19 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Number of symptomatic patients affected by COVID-19 | 7-60 days after the 2nd dose of vaccine
  Evaluating the protection conferred by vaccination, by detecting the number of symptomatic pts affected by COV, diagnosed 7-60 days after the 2nddose of vaccine. Confirmed of COV infection is defined according to the Food and Drug Administration criteria combined with a nasopharyngeal swab, positive for SARS-Cov-2, obtained during the symptomatic period or within 4 days before or after it.

SECONDARY OUTCOMES:
Antibodies variation at different timepoints | baseline and 30(±7), 180(±7),365(±7)days after the 2nd dose of vaccine
  Two tests are used: LIAISON SARS-Cov-2 TrimericSIgG and Elecsys anti-SARS-Cov-2; The combined use of the two dosages in this vaccinated population will allow an assessment of the pre-vaccine immunological status and the characterization of the antibodies produced after the vaccination stimulus
Adverse Events and interference between vaccine and cancer treatments | from 7 to 90 days after the 2nd dose of vaccine
  collection of AEs in a paper form completed by patients

CONTACTS AND LOCATIONS:
Overall Officials: MARGHERITA RATTI, MD, Principal Investigator — Azienda Socio Sanitaria Territoriale di Cremona (ASST Cremona)
Locations (1):
- UO Oncologia, ASST di Cremona, Cremona, Lombardy, Italy